CLINICAL TRIAL: NCT05627973
Title: Health Status of < 50 Year Old Patients After Surgically Implanted Biological and Mechanical Aortic Valves: a Population-based Retrospective Analysis (2010-2020)
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Sicknessfund Burgenland (Unknown); Landesklinikum Sankt Polten (Other)
Responsible Party: Principal Investigator, Hendrik Jan Ankersmit, Univ. Prof. , MD, MBA, Medical University of Vienna
Other Study IDs: AUTHEARTVISIT < 50
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Aortic valve replacement with mechanical valves
  Interventions: Device: Aortic Valve Replacement
- Aortic valve replacement with bioprostheses
  Interventions: Device: Aortic Valve Replacement

INTERVENTIONS:
Device: Aortic Valve Replacement — Surgical replacement of aortic valves

SUMMARY:
The overall project aim is to study outcomes following aortic valve replacement with either mechanical valves or bioprostheses by retrieving data from the main social security carriers in Austria for the years 2010-2020 in under 50 year old patients.

DETAILED DESCRIPTION:
The purpose of this research project is to evaluate mortality (primary outcome) and incidence of heart attack, stroke, reoperation and first diagnosis of heart insufficiency, MACE (secondary outcomes) after aortic valve replacement in under 50 year olds. We aim to compare those outcomes between mechanical valves and bioprostheses.

Data will be retrieved from the main social security carriers in Austria (covering 98% of its population) from 2010-2020.

ELIGIBILITY:
Inclusion Criteria:

* isolated surgical aortic valve replacement in Austria

Exclusion Criteria:

* below 18 years of age
* above 50 years of age
* concomitant heart surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients who underwent isolated surgical aortic valve replacement in Austria above 18 years and below 50 years of age with no other concomitant heart surgery were included.
Sampling Method: Non-Probability Sample
Enrollment: 991 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Overall mortality | 10 years
  all cause mortality after aortic valve replacement

SECONDARY OUTCOMES:
reoperation | 10 years
  incidence of reoperation after aortic valve replacement
stroke | 10 years
  incidence of stroke after aortic valve replacement
heart attack | 10 years
  incidence of heart attack after aortic valve replacement
heart insufficiency | 10 years
  incidence of heart insufficiency after aortic valve replacement
MACE | 10 years
  incidence of MACE after aortic valve replacement

IPD SHARING:
Plan to Share IPD: No